CLINICAL TRIAL: NCT03317561
Title: Etiology of Myocardial Injury Following Non-cardiac Surgery - a Prospective Clinical Trial
Brief Title: Myocardial Injury Following Non-cardiac Surgery
Acronym: EMINENT
Status: Completed | Type: Observational
Sponsor: Karolinska Institutet (Other)
Collaborators: Karolinska University Hospital (Other)
Responsible Party: Principal Investigator, Anil Gupta, Associate Professor, Karolinska Institutet
Other Study IDs: 2017-11-01
Record Dates: First submitted 2017-10-18; First posted 2017-10-23 (Actual); Last update posted 2023-10-05 (Actual); Status verified 2023-10

CONDITIONS: Myocardial Injury; Surgery--Complications
Keywords: troponin; major surgery

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — Plasma
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Myocardial injury: Subjects who have had an increase in troponin T level (> 99 percentile) in the perioperative period shall form the cases.
- Control: Subjects who do not have an increase in troponin T level (< 99 percentile) in the perioperative period shall form the controls.

SUMMARY:
It is estimated that > 200 million patients in the world undergo surgery each year of which approximately 10 million will suffer from a myocardial injury in the perioperative period. Mortality is high in patients with myocardial injury since it often goes undiagnosed and management is unclear. In contrast to myocardial infarction diagnosed in the emergency room (non-surgical patient) where treatment is well established today, patients suffering from a perioperative myocardial injury have a poorer outcome. Additionally, the patho-physiology of myocardial injury is unknown in the individual patient, non-invasive diagnostic tools are not widely available and treatment remains unknown.

Most cases of myocardial injury in Non-cardiac surgery (MINS) are seen within the first 48-72 h after surgery and a majority have no symptoms. Many patients developing MINS are < 65 years old and non-diabetics, an age group that usually does not have coronary artery disease. A elevated Troponin T (TnT) without symptoms or ECG changes, typically occurring in the perioperative period, is an independent predictor of 30-day mortality. Surgical trauma also causes an increase in several pro-inflammatory cytokines, which together with sympathetic over-activity and platelet activation, leads to a hyper-coagulant state, and in turn may cause coronary thrombosis. It is possible that some cases of MINS also result from oxygen supply-delivery mismatch. To our knowledge, no study has investigated the cause of MINS in patients presenting with increased TnT in the perioperative period. Our aim is therefore to investigate patients having MINS in order to better understand its aetiology and subsequently develop focused strategies to reduce risks.

DETAILED DESCRIPTION:
Introduction:

It is estimated that > 200 million patients in the world undergo surgery each year of which approximately 10 million would suffer from a myocardial injury in the perioperative period. Mortality is high in this group of patients since it often goes undiagnosed, the patho-physiology of myocardial injury is unclear, non-invasive diagnostic tools are not widely available and treatment is unknown.

Multiple studies have shown that > 10% of patients > 65 years and undergoing non-cardiac surgery have an increase in Troponin T (TnT). In the POISE study including 8331 patients, the authors found that 5.7% of the placebo group suffered from a myocardial injury within the 30-day postoperative period. In the recently published data from the VISION study including > 15,000 patients, the authors demonstrated that patients with peak perioperative TnT values of < 0.01, 0.02, 0.03-0.29 and > 0.30 ng/L had a 30-day mortality of 1%, 4%, 9.3% and 16.9% respectively. Furthermore, an elevated TnT without symptoms or ECG changes are an independent predictor of 30-day mortality. It is possible that some cases of myocardial injury in Non-cardiac surgery (MINS) result from oxygen supply-delivery mismatch due to severe perioperative hypotension, and possibly persistent tachycardia but coronary artery thrombosis cannot be excluded in these patients. It is well known that surgical trauma causes an increase in several pro-inflammatory cytokines which, together with sympathetic over-activity, leads to a hypercoagulable state due to platelet activation, and a predisposition to thrombosis. In one study, it was found that approximately 1/3 of the patients had evidence of intracoronary thrombosis at autopsy.

Myocardial infarction with non-obstructive coronary artery (MINCA) has recently received greater attention in the literature. The underlying patho-physiology responsible for MINCA revealed the presence of a typical myocardial infarct on cardiac magnetic resonance imaging in only 24% of patients, with myocarditis occurring in 33% and no significant abnormality in 26%. A rare cause of MINCA is Takotsubo cardiomyopathy, also called stress cardiomyopathy. Recently, coronary angiography using computerized tomographic angiography (CTA) has added a new dimension to the diagnostic armamentarium available to the clinician. Using advanced imaging techniques and low radiation, it is today possible to determine quite accurately coronary artery anatomy and thereby determine stenotic lesions in the coronary vasculature. Echocardiography can be easily performed by an experienced technician, the images stored digitally and evaluated subsequently by specialists. The availability of continuous perioperative monitoring of several hemodynamic indices as well as regular blood gas analysis, may enable determination of oxygen demand-supply mismatch.

Methods:

This is a case-control study in patients undergoing major, non-cardiac surgery. Permission will be obtained from the Ethics committee prior to patient recruitment and Good Clinical Practice guidelines will be followed in all patients. Two parts to the study are planned:

Part 1. Screening of all patients undergoing vascular surgery (arterial surgery) where demographic data, co-morbidities, laboratory and perioperative haemodynamic parameters, postoperative complications will be recorded and patients followed up at 30, 90 and 365 days after surgery via medical records. This group is estimated to include 500 patients. Informed consent will be obtained from these patients for data collection and follow-up via medical records.

Part 2. Patients with a significant increase in TnT (estimated 10% = 50 patients) will undergo cMRI (see below) and a matched control without increase in TnT will also undergo similar protocol as described below.

Verbal and written informed consent will be obtained from all patients willing to participate in the second part of the study. The following laboratory tests would be performed preoperatively (baseline values): routine bloods, creatinine, urea, estimated glomerular filtration rate (eGFR), C-reacting proteins (CRP), white blood cell (WBC) count, TnT, N-Terminal pro-Brain Natriuretic Peptide (NT-pro BNP), lipid profile, 12-lead EKG and echocardiography (ECHO).

Anaesthesia and Surgery The surgical and anaesthetic techniques would be determined by physicians responsible for the patient and according to established hospital routines and practices. Patient records would be used for the determination of adverse events according to a standardized protocol. Patient characteristics, pre-operative risk factors, laboratory data and follow-up data would be obtained from medical records. Prophylaxis against deep vein thrombosis, surgical infections and fluid and electrolyte balance would also follow hospital practice. All included patients would be admitted to the post-anaesthesia care unit (PACU) overnight, and longer if deemed necessary by the attending Anaesthesiologist. Patients would be continuously haemodynamically monitored and anaesthesia records would be maintained for independent assessment by a blinded reviewer. Drop in blood pressure that persists despite short-acting vasopressors will be treated by infusion of noradrenaline perioperatively. Hs-TnT would be repeated in all patients at 24, 48 and 72 h postoperatively. Plasma NT-pro BNP would be re-assessed at 24 h. A 12-lead EKG would be recorded in all patients with elevated high-sensitivity TnT (hs-TnT) at the time of first occurrence and 48 h later. Platelet function tests, microparticles as well as coagulation tests would be performed periodically in the perioperative period. Further laboratory tests would be performed as needed at the discretion of the attending physician.

Cardiac Magnetic Resonance Imaging (cMRI) would be performed within 1-3 days of detecting a rise in TnT in the study population as well as the control group. This will include a drug-induced (Adenosine) stress test of the heart in connection with the examination. cMRI will allow an increased opportunity to identify an acute myocardial injury, even of a minor nature, and minimises the risk of radiation to patients (as with CTA). The cMRI scan will be performed within 24-48 hours after elevated levels of cTnT (cardiac troponins) are measured.

Echocardiography: Protocolized ECHO would be performed 24 h after detection of raised TnT in the study group, and at corresponding time period in a matched group of controls. The ECHO will be recorded and subsequently interpreted by an experienced clinical physiologist/cardiologist to determine wall motion abnormalities and systolic and diastolic function.

When deemed necessary by the attending Cardiologist, the following may also be performed:

Conventional invasive coronary angiography: This will only be done at the discretion of the attending Cardiologist and in agreement with the patient and surgeon at an appropriate time point after surgery, if deemed necessary.

The control group will be matched for age, sex and co-morbidities described in the revised cardiac risk score (myocardial ischemia, cardiac failure, stroke, diabetes mellitus, renal insufficiency and major-risk surgery) (ref) and grouped into < 3 risk factors and >/= 3 risk factors.

ELIGIBILITY:
Inclusion Criteria:

1. Patients in the age group > 45 years
2. Non-cardiac, vascular surgery

Exclusion Criteria:

1. Patients with atrial fibrillation
2. Moderate-severe renal insufficiency (GFR < 50)
3. Allergy to iv contrast or drugs used for diagnostics will be excluded
4. Known lung embolism
5. Inability to comprehend the study or language barriers

Ages: 45 Years to 100 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with an increase in Troponin T (> 20 ng/L) or a > 50% rise from preoperative values after induction of anesthesia will form the Myocardial injury Group while those without an increase in Troponin T (< 14 ng/L) will form the Control group
Sampling Method: Non-Probability Sample
Enrollment: 450 (Actual)
Dates: Start 2017-12-01 (Actual); Primary Completion 2023-03-31 (Actual); Study Completion 2023-06-30 (Actual)

PRIMARY OUTCOMES:
Myocardial injury as seen by cMRI | < 3 days after rise in Troponin T
  Number of patients with a significant myocardial detected by cMRI in relation to the number that had an increase in TnT postoperatively

SECONDARY OUTCOMES:
Protocolized echocardiography | < 48 hours after rise in Troponin T
  Number of patients with wall motion abnormalities and systolic and diastolic function as assessed by a competent person.
Kidney injury | < 3 days after induction of anesthesia
  Number of patients with a significant increase in creatinine postoperatively as determined by the KIDCO criteria
Mortality | Within 365 days
  The number of patients that have an increase in TnT and die at 30, 90 and 365 days in relation to those who have normal values
Number of patients with significant Hypotension (perioperative) | 24 hours after induction of anesthesia
  Average perioperative direct arterial blood pressures (systolic, mean, diastolic measured in mmHg) will be compared in groups with raised TnT and normal TnT
Number of patients with significant ST-T segment changes (perioperative) | 0 - 24 hours anesthesia induction
  Electronic determination of significant changes in ST-T segment analysed continuously determined using hexad on a Philips monitoring system

CONTACTS AND LOCATIONS:
Overall Officials: Anil Gupta, MD, PhD, Principal Investigator — Department of Clinical Research, and PMI, Karolinska Hospital
Locations (1):
- Karolinska Hospital, Solna, Stockholm, Sweden

IPD SHARING:
Plan to Share IPD: No
Not planned as of today

REFERENCES:
- [Derived] Valadkhani A, Gupta A, Cauli G, Nordstrom JL, Rohi A, Tufexis P, Hallsjo Sander C, Jacobsson M, Bell M. Diastolic Versus Systolic or Mean Intraoperative Hypotension as Predictive of Perioperative Myocardial Injury in a White-Box Machine-Learning Model. Anesth Analg. 2025 Jul 1;141(1):5-15. doi: 10.1213/ANE.0000000000007379. Epub 2025 Feb 20. PMID 39977341